CLINICAL TRIAL: NCT02382588
Title: A Prospective, Double-masked, Placebo Controlled Comparison of Topical 0.15% Gancyclovir Gel (Zirgan) Versus 0.3% Hypromellose Gel (Genteal Gel; Placebo) for the Treatment of Herpes Zoster Keratitis
Brief Title: Comparison of Topical 0.15% Gancyclovir Gel Versus 0.3% Hypromellose Gel for the Treatment of Herpes Zoster Keratitis
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: There were difficulties meeting the enrollment goal within stipulated time frames.
Sponsor: Northwestern University (Other)
Collaborators: Bausch & Lomb Incorporated (Industry)
Responsible Party: Principal Investigator, Robert Feder, Professor of Ophthalmology, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4321
Record Dates: First submitted 2015-03-03; First posted 2015-03-06 (Estimated); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-06

CONDITIONS: Herpes Zoster Keratitis
MeSH Terms: interventions — Ganciclovir

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gancyclovir gel (Experimental): 0.15% gancyclovir gel to be applied in the affected eye 5 times per day for a week, followed by 3 times per day for an additional 7 days or until the healing of the dendrite, whichever is earlier.
  Interventions: Drug: gancyclovir gel
- hypromellose gel (Placebo Comparator): 0.3% hypromellose gel to be applied in the affected eye 5 times per day for a week, followed by 3 times per day for an additional 7 days.
  Interventions: Drug: Hypromellose gel

INTERVENTIONS:
Drug: gancyclovir gel — 0.15% gancyclovir gel to be applied in the affected eye 5 times per day for a week, followed by 3 times per day for an additional 7 days or until the healing of the dendrite, whichever is earlier.
  Other Names: zirgan
  Arms: Gancyclovir gel
Drug: Hypromellose gel — 0.3% hypromellose gel to be applied in the affected eye 5 times per day for a week, followed by 3 times per day for an additional 7 days.
  Other Names: genteal gel
  Arms: hypromellose gel

SUMMARY:
The purpose of this study is to evaluate the efficiency of topical gancyclovir 0.15% in the treatment of herpes zoster keratitis. Half the patients will receive the study drug while the other half of the patients will receive the placebo

DETAILED DESCRIPTION:
Patients with herpes zoster keratitis will be enrolled in the study. All patients will receive oral anti-viral medication as a standard-of-care therapy. The patients will be randomized into two groups and given either the study drug or the placebo at the time of enrollment. The patients will come for weekly visits during which slit lamp photograph of the dendrite will be taken. At week 2, if the dendrite has not healed the drug will by unmasked and rescue therapy will be given. the patients will be examined at week 1, 2, and 3 or until resolution occurs.

ELIGIBILITY:
Inclusion Criteria:

* age 18 and above
* have not been on gancyclovir gel or any other form of topical antiviral therapy for the past month
* able and willing to attend subsequent follow-up visits

Exclusion Criteria:

* Associated retinitis
* patients who are allergic to gancyclovir
* patients who will require systemic or intra-vitreal gancyclovir therapy
* patients who are pregnant or breastfeeding

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-12-10 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwestern University, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Once the study is completed study results will be shared with the study subjects.

REFERENCES:
- [Background] Liesegang TJ. Herpes zoster ophthalmicus natural history, risk factors, clinical presentation, and morbidity. Ophthalmology. 2008 Feb;115(2 Suppl):S3-12. doi: 10.1016/j.ophtha.2007.10.009. PMID 18243930
- [Background] Ostler HB, Thygeson P. The ocular manifestations of herpes zoster, varicella, infectious mononucleosis, and cytomegalovirus disease. Surv Ophthalmol. 1976 Sep-Oct;21(2):148-59. doi: 10.1016/0039-6257(76)90092-8. PMID 185734
- [Background] Liesegang TJ. Corneal complications from herpes zoster ophthalmicus. Ophthalmology. 1985 Mar;92(3):316-24. doi: 10.1016/s0161-6420(85)34034-4. PMID 3873048
- [Background] Trousdale MD, Nesburn AB, Willey DE, Taaid H. Efficacy of BW759 (9-[[2-hydroxy-1(hydroxymethyl)ethoxy]methyl]guanine) against herpes simplex virus type 1 keratitis in rabbits. Curr Eye Res. 1984 Aug;3(8):1007-15. doi: 10.3109/02713688409011747. PMID 6333319
- [Background] Villarreal EC. Current and potential therapies for the treatment of herpes-virus infections. Prog Drug Res. 2003;60:263-307. doi: 10.1007/978-3-0348-8012-1_8. PMID 12790345

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Per review of consent and drug diaries, 8 subjects were enrolled.
Period: Overall Study
Arm/Group | Gancyclovir Gel | Hypromellose Gel
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Report on "Comparison of Topical 0.15% Gancicyclovir Gel vs 0.3% Hypromellose Gel for the treatment of Herpes Zoster keratitis
  This study was begun in December of 2013 in order to determine if topical ganciclovir 0.15% was beneficial in the treatment of Herpes Zoster keratitis. Despite the number of years the study was open we were only able to recruit 8 subjects. Data was not summarized due to privacy concerns for participants due to low enrollment The study was closed in May of 2020.
Groups:
- Total: Total of all reporting groups
Arm/Group | Gancyclovir Gel | Hypromellose Gel | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 8
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 4 | 3 | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Corneal Ulcer Healing
Description: Based on weekly slitlamp photographs
Time Frame: 2 weeks
Population: as for baseline characteristics
Arm/Group | Gancyclovir Gel | Hypromellose Gel
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Throughout each patient's participation. 4 visits throughout a maximum of 2 months.
Description: Report on "Comparison of Topical 0.15% Gancicyclovir Gel vs 0.3% Hypromellose Gel for the treatment of Herpes Zoster keratitis
  This study was begun in December of 2013 in order to determine if topical ganciclovir 0.15% was beneficial in the treatment of Herpes Zoster keratitis. Unfortunately despite the number of years the study was open we were only able to recruit 7 subjects into the study. This was not enough to provide meaningful results. The study was closed in May of 2020.
Arm/Group | Gancyclovir Gel | Hypromellose Gel
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/88/NCT02382588/Prot_SAP_000.pdf